CLINICAL TRIAL: NCT06778603
Title: Resection of Osteosarcoma in Limbs Navigated by B7H3-based NIR Lmaging: a Prospective, Single-center,Single-arm, Exploratory Trial
Brief Title: B7-H3 NIR Imaging for Osteosarcoma Surgery
Acronym: ROLN-B7-H3
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Simcere Pharmaceutical Group Limited (Unknown)
Responsible Party: Principal Investigator, Xie Lu, Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 22
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Osteosarcoma; Resection Margins; B7-H3 Probe; Local Recurrence
Keywords: osteosarcoma; resection margins; B7-H3 Targeted Probe; local recurrence rate
MeSH Terms: conditions — Osteosarcoma; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Drug: a targeted probe B7H3-IRDye800CW

INTERVENTIONS:
Drug: a targeted probe B7H3-IRDye800CW — B7H3-IRDye800CW was synthesized by conjugating IRDye800CW NHS Ester and Anti-B7H3 antibody.

SUMMARY:
Complete removal of all tumor tissue with a wide surgical margin is essential for the treatment of osteosarcoma (OS). However, it's difficult, sometimes impossible, to achieve due to the invisible small satellite lesions and blurry tumor boundaries. Besides, intraoperative frozen-section analysis of resection margins of OS is often restricted by the hard tissues around OS, which makes it impossible to know whether a negative margin is achieved. Herein, based on the high expression of B7-H3 in OS, a targeted probe B7H3-IRDye800CW is synthesized by conjugating anti-B7H3 antibody and IRDye800CW. This trial is aimed to investigate R0-resection rate and 2-y local recurrence rate after using this probe in Musculoskeletal tumor surgery for osteosarcoma as well as the safety parameters of this probe in human.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with histologically confirmed osteosarcoma of the limbs.
* 2. the patients has not undergone tumor resection.
* 3. Age between 18 and 60 years old.
* 4. No prior systemic treatment for osteosarcoma.
* 5. Measurable disease as assessed by imaging studies (e.g., MRI, CT).
* 6. Adequate bone marrow, liver, and renal function.
* 7. Written informed consent obtained from the patient.

Exclusion Criteria:

* 1. History of other malignancies within the past 5 years.
* 2. Pregnancy or lactation.
* 3. Known hypersensitivity to any component of the B7H3-based NIR imaging agent.
* 4. Uncontrolled intercurrent illness that would preclude safe study participation.
* 5. Prior radiation therapy to the target lesion.
* 6. Any medical condition that would compromise the patient's ability to undergo surgery or comply with study procedures.
* 7.Patients not able to sign the Informed Consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 21 days
  According to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Musculoskeletal Tumor Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng F, Li C, Wang H, Wang Y, Ren T, He F, Jiang J, Xu J, Wang B, Wu Y, Yu Y, Hu Z, Tian J, Wang S, Tang X. Intraoperative Resection Guidance and Rapid Pathological Diagnosis of Osteosarcoma using B7H3 Targeted Probe under NIR-II Fluorescence Imaging. Adv Sci (Weinh). 2024 Sep;11(33):e2310167. doi: 10.1002/advs.202310167. Epub 2024 Mar 19. PMID 38502871